CLINICAL TRIAL: NCT02446522
Title: Comparative Results of Endoscopic and Open Methods of Vein Harvesting for Coronary Artery Bypass Grafting: a Prospective Randomized Parallel-group Trial.
Brief Title: Compare Endoscopic and Open Methods of Vein Harvesting for Coronary Artery Bypass Grafting
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EVH vs OVH
Record Dates: First submitted 2015-05-13; First posted 2015-05-18 (Estimated); Last update posted 2015-05-18 (Estimated); Status verified 2015-05

CONDITIONS: Autovenous Conduit for Coronary Artery Bypass Grafting

ARMS (2):
- Open vein harvesting (Active Comparator): Patients with IHD, who were underwent open vein harvest method (OVH)
  Interventions: Procedure: Open vein harvesting
- Endoscopic vein harvesting (Active Comparator): Patients with IHD, who were underwent edoscopic vein harvestingopen vein harvest method (EVH).
  Interventions: Procedure: Endoscopic vein harvesting

INTERVENTIONS:
Procedure: Open vein harvesting — Open vein harvesting was performed as a continuous incision under vision control. The GSV was identified two fingers proximal to the medial malleolus according to the standard practice. The vein was harvested using Metzenbaum scissors, and a continuous incision was made along the route of the vein. Care was taken not to traumatize the nerve, vein or its branches. Vein branches were ligated with titanium clips. The wound was closed in layers with continuous 2-0 Polysorb sutures and 3-0 skin sutures.
  Arms: Open vein harvesting
Procedure: Endoscopic vein harvesting — Endoscopic vein harvesting was performed through minimal incisions with use of Vasoview 6 system (Maquet Medical Systems, Wayne, NJ, USA.) The vein was identified through a 3 cm incision below the knee. The incision site was sealed using a balloon port to create a tunnel inside the leg. A second unit with cautery was inserted via the port to cut and seal the tributary branches. A 1 cm skin incision was made near the groin to ligate the distal end of the GSV and remove the vein, which was checked for leakage. The wound was closed with 3-0 skin sutures
  Arms: Endoscopic vein harvesting

SUMMARY:
There is no shared vision relating to integrity and quality of the conduit after the impact on the vein wall during vein harvesting. In this connection, the investigators studied the initial state of the venous conduit, interoperation damages of the vein and postoperative wound complications while using two methods of GSV harvesting.

DETAILED DESCRIPTION:
The great saphenous vein (GSV) remains one of the most commonly used conduits due to its ease of harvest, availability and versatility [1] Traditional harvesting of GSV is open vein harvesting, which involves an extended leg incision. This technique is associated with a significant morbidity and wound complications occur in 2-24% of cases.

Minimally invasive techniques endoscopic vein harvesting (EVH), have therefore been developed to reduce post-CABG leg wound complications. Last time the endoscopic vein harvesting is the method of choice in many centers as it allowed reduction of post-surgical complications as compared to the open method. Although long-term graft patency following EVH has been questioned cohort studies have reported that the technique is safe and effective.

The possibility to use lymphoscintigraphy for evaluation of lower limb lymphatic system after vein harvesting for the coronary artery bypass surgeries was reported before. Nevertheless, the state of the lymphatic system after vein harvesting remains to be poorly studied.

Currently, there is no shared vision relating to integrity and quality of the conduit after the impact on the vein wall during vein harvesting. In this connection, the investigators studied the initial state of the venous conduit, interoperation damages of the vein and postoperative wound complications while using two methods of GSV harvesting.

ELIGIBILITY:
Inclusion Criteria:

* subjects with multivascular lesion of the coronary artery to whom coronary artery bypass surgery was indicated.

Exclusion Criteria:

* urgent coronary artery bypass surgery with unstable haemodynamics;
* previous coronary artery bypass surgery;
* chronic venous insufficiency С4-С6 under СЕAR classification;
* previous limb surgeries.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2010-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
postoperative wound complications | during 30 day after operation
  all cases postoperative wound complications